CLINICAL TRIAL: NCT04496310
Title: Telemedicine With Mobile Internet Devices for Innovative Care of Patients With Epilepsy
Brief Title: Tele-epic (Telemedicine for Epilepsy Care)
Acronym: Tele-epic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Usl di Bologna (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GR-2018-12365475
Record Dates: First submitted 2020-07-06; First posted 2020-08-03 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Epilepsy; Epileptic Encephalopathy; Refractory Epilepsy
Keywords: Telemedicine; Epilepsy; Antiepileptic drugs monitoring
MeSH Terms: conditions — Epilepsy; Drug Resistant Epilepsy | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine (Experimental): Baseline: in office clinical assessment of all patients (collection of seizure diary).
  Followup: scheduled 6-month consultations through a telemedicine device providing remote outcome assessment, counselling and follow-up. If required, on call video consultations available by contacting a provider through telemedicine, 3-hr/week.
  Interventions: Procedure: Telemedicine
- Usual care (No Intervention): Baseline: in office clinical assessment of all patients (collection of seizure diary).
  Followup: scheduled 6-month in-office consultations with outcome assessment, counselling and follow-up. On-call consultations are possible if needed by the patient, by contacting a clinician through an in-office phone call, 3-hr/week.

INTERVENTIONS:
Procedure: Telemedicine — Telemedicine versus usual care (face to face visit)
  Arms: Telemedicine

SUMMARY:
Epilepsy is a chronic condition that requires consistent follow-up aimed at seizure control, surveillance of comorbidities, monitoring of antiepileptic drugs (AED) levels and side effects. Patients may encounter difficulties to be assessed adequately and the disease burden is increased by the need for travelling across the country for medical consultations. Driving restrictions are a further limit to access specialized Centers able to provide an integrated approach focused on patient needs. Telemedicine (TM) offers an invaluable support to patient follow-up, joining the sparse distribution of patients in the country with the prompt availability of a team of experts. The project assesses, through a randomized controlled trial, the non-inferiority of TM in monitoring seizure control compared to usual (face-to-face) care. This approach, coupled with a new self home-sampling method for the measurement of AED levels, will reduce health care costs and simplify patients management.

ELIGIBILITY:
Inclusion Criteria:

* adult (age>18 yrs) and pediatric (age<18yrs) outpatients with established diagnosis of epilepsy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-07-09 (Actual); Primary Completion 2023-07-08 (Estimated); Study Completion 2023-07-08 (Estimated)

PRIMARY OUTCOMES:
Seizures control through seizure diary | 3 years
  Non-inferiority in seizures control of follow-up procedures through video consultations with telemedicine devices versus in-office, usual care (UC).
  Outcomes: non-inferiority of mTM on the primary end-point (seizure control assessed through seizure diary) at 18 month follow- up.
  Assessment of "seizure control" at the end of 18 month-follow-up. Clinical worsening defined as at least 1: (i) fall of at least 2 positions of the following frequency categories: daily/multiple per day; multiple/week, weekly; multiple/month; monthly; multiple/year; annual; (ii) relapse after SF; (iii) new-onset/relapse of convulsive seizures, tonic/atonic seizures with fall, status epilepticus.

SECONDARY OUTCOMES:
Adherence to treatment | 3 years
  Comparing Adherence to treatment (trough anti epileptic drug monitoring) among telemdicne group and usual care group
ADRs - Adverse Events Profile-AEP | 3 years
  Comparing adverse drugs reactions among telemdicne group and usual care group (Adverse Events Profile-AEP)
Quality of life (QoL) | 3 years
  Comparing quality of life among telemdicne group and usual care group (QoL In Epilepsy-QOLIE- 31,1.0,)
Pediatric quality of life (PedsQL) | 3 years
  Comparing pediatric quality of life among telemdicne group and usual care group (Pediatric QoL Inventory-PedsQL)
Mood-disorders - Beck Depression | 3 years
  Comparing the occurence of mood-disorders (Beck Depression Inventory-BDI-II)
Mood-disorders - State-Trait Anxiety | 3 years
  Comparing the occurence of mood-disorders (State-Trait Anxiety Inventory-STAI Y-1,2)
Mood-disorders - Child Behavior | 3 years
  Comparing the occurence of mood-disorders (Child Behavior CheckList-CBCL for patients aged 6-18 yrs)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda USL di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Licchetta L, Trivisano M, Baldin E, Mohamed S, Raschi E, Mostacci B, Zenesini C, Contin M, Vigevano F, Bisulli F, Tinuper P, Vignatelli L. TELEmedicine for EPIlepsy Care (TELE-EPIC): protocol of a randomised, open controlled non-inferiority clinical trial. BMJ Open. 2021 Dec 3;11(12):e053980. doi: 10.1136/bmjopen-2021-053980. PMID 34862297